CLINICAL TRIAL: NCT07168265
Title: The Effects of Androgen Replacement Therapy on Tear Osmolarity and Ocular Surface Parameters in Androgen Deficiency
Acronym: EffAndonOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neon Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMU KAEK 2021/557; OMU (Other: Ondokuz Mayıs University)
Record Dates: First submitted 2025-06-21; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Androgen Deficiency; Ocular Surface Disease; Tear Osmolarity
Keywords: androgen deficiency; ocular surface; tear osmolarity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- testosterone (Other)
  Interventions: Drug: androgen replacement therapy

INTERVENTIONS:
Drug: androgen replacement therapy — intramuscular testosterone

SUMMARY:
Objective: To evaluate tear osmolarity and ocular surface findings in men with androgen deficiency (AD) and assess changes after androgen replacement therapy (ART).

Design: A prospective interventional study. Participants and Methods Right eyes of 77 male participants were evaluated in this study. Serum total testosterone level were measured, and participants were categorized as AD group (testicular hypofunction, n=37, testosterone level <231 ng/dL) and control group (healthy controls, n=40, testosterone level >346 ng/dL). The parameters including Aging Male Symptoms Scale(AMS), OSDI scores, Meibomian Gland Dysfunction- Grading System(MGD-GS) scores, corneal staining, tear break-up time(TBUT), Schirmer I/II tests, tear osmolarity, the depth (TMD), the height (TMH) and the area (TMA) of inferior tear meniscus were investigated. AD group received intramuscular testosterone every two weeks.

Main Outcome Measures: The changes in the ocular surface parameters were investigated during the ART while comparing the values of these parameters between the AD and control groups at baseline, 6th and 18th weeks of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Androgen deficiency

Exclusion Criteria:

* having any ocular disease, history of surgery, drop use

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Tear Osmolarity in mOsm/L | 5 months
  Tear osmolarity was measured by TearLab device in patients. The changes in the tear osmolarity were investigated during the ART while comparing the values of these parameters between the AD and control groups at baseline, 6th and 18th weeks of the treatment.
Schirmer Test in mm | 5 months
  Schirmer Test is applied by Schirmer tear paper after anesthesic drop administration into the eye.
Tear break-up time (TBUT) in sec | 5 months
  TBUT is measured by ophthalmologist after application of fluorecein dye.
MGD-GS score in number | 5 months
  MGD-GS score was performed by ophthalmolgist using biomicroscopy
Questionary Scoring in number | 5 months
  AMS and OSDI scoring charts were completed by the participants.
Optical Coherence Tomography findings: TMH, TMA, and TMD in microns | 5 months
  Tear meniscus height (TMH), area (TMA), and depth (TMD) were measured by Optical coherence tomography in each participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)